CLINICAL TRIAL: NCT00400218
Title: Evaluate the Safety and Tolerability of Hyzaar(R) (Losartan 50 Mg/ Hydrochlorothiazide 12.5 Mg) In the Treatment of Hypertension
Brief Title: Evaluate the Safety and Anti-Hypertensive Efficacy of Hyzaar(R) In Patients With Mild To Moderate Essential Hypertension (0954A-323)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0954A-323; 2006_049
Record Dates: First submitted 2006-11-15; First posted 2006-11-16 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Hydrochlorothiazide; Losartan; Duration of Therapy

INTERVENTIONS:
Drug: MK0954A, hydrochlorothiazide (+) losartan potassium / Duration of Treatment: 12 Weeks

SUMMARY:
Evaluate the safety and anti-hypertensive efficacy of hyzaar(R) in patients with mild to moderate essential hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Patient is either receiving high blood pressure monotherapy or no treatment
* Patient will have reached the legal age by the time enter the study
* Patients diagnosed with mild to moderate essential high blood pressure or high blood pressure with other conditions such as diabetes or cardiovascular diseases and are taking high blood pressure medication (exclude diuretic), but did not meet treatment goal

Exclusion Criteria:

* Patient with high levels of uric acid in the blood who has received medications for uric acid in the urine within 3 months prior to enrollment
* Patients who are hypersensitive to any component of the study medication
* Patients who are hypersensitive to other sulfonamide-derived drugs
* Patients with anuria (hyzaar(R) is not recommended for patients with hepatic impairment or severe renal impairment, creatinine clearance </= 30 ml/min)
* Unstable diabetes (hba1c > 8%), or a change in diabetes medication during study treatment. patients with stable diabetes may enter the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2005-09-01 (Actual); Primary Completion 2006-07-01 (Actual); Study Completion 2006-07-19 (Actual)

PRIMARY OUTCOMES:
Blood pressure over 12 weeks
Safety and Tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC